CLINICAL TRIAL: NCT02741661
Title: Determinants of Coronary Tortuosity
Brief Title: Influence of Myocardial Shortening on Coronary Tortuosity
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jonathan R. Lindner, MD, Professor, Oregon Health and Science University
Other Study IDs: Coronary Tortuosity
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Coronary Artery Vessels; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal coronary arteries: Patients in whom coronary arteriography has demonstrated no significant tortuosity.
  Interventions: Other: No intervention. Observational study
- Tortuous coronary arteries: Patients in whom coronary arteriography has demonstrated tortuous coronary arteries defined as >1 major bend of >45 degrees in a major coronary artery
  Interventions: Other: No intervention. Observational study

INTERVENTIONS:
Other: No intervention. Observational study — No intervention

SUMMARY:
This study is a retrospective analysis where coronary arteriograms are being analyzed to determine whether the presence of tortuous coronary arteries correlate with any specific measures of left ventricular mass or left ventricular function on echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* subjects referred for angiography
* echocardiography performed within 3 months.

Exclusion Criteria:

* connective tissue disease
* severe LV dysfunction
* prior coronary artery bypass surgery
* major adverse coronary event between angiogram and echo procedures
* moderate or greater valve disease
* acute coronary syndrome

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective study of subjects who have undergone clinically-indicated coronary arteriography who also have an echocardiogram that was performed within 3 months of the angiogram.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2015-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Degree of longitudinal shortening | 3 months
  Measurement of longitudinal shortening of the left ventricle measured on an echocardiography (retrospectively) that was performed within 3 months of the angiogram

SECONDARY OUTCOMES:
LV mass | 3 months
  Measurement of longitudinal shortening of the left ventricle measured on an echocardiography (retrospectively) that was performed within 3 months of the angiogram

CONTACTS AND LOCATIONS:
Locations (1):
- OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes